CLINICAL TRIAL: NCT05190393
Title: Comparison of Techniques Between Concave Distraction and Convex Resection in the Treatment of Congenital Cervical Scoliosis
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUTHCCS
Record Dates: First submitted 2021-12-06; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2016-01

CONDITIONS: Congenital Scoliosis Due to Bony Malformation; Cervical Scoliosis
Keywords: Congenital cervical scoliosis; hemivertebra resection; distraction and lateral opening; spinal fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Convex resection group: Patients were used hemivertebra resection procedure on convex side to treat congenital cervical scoliosis.
  Interventions: Procedure: hemivertebra resection on convex side
- Concave distraction group: Patients were used distraction and lateral opening procedure on concave side to treat congenital cervical scoliosis, without hemivertebra resection.
  Interventions: Procedure: concave distraction group

INTERVENTIONS:
Procedure: hemivertebra resection on convex side — Patients were used hemivertebra resection procedure to treat congenital cervical scoliosis.
  Groups: Convex resection group
Procedure: concave distraction group — Patients were used distraction and lateral opening procedure to treat congenital cervical scoliosis.
  Groups: Concave distraction group

SUMMARY:
To treat congenital cervical scoliosis, previous literature introduced surgical technique, like hemivertebra resection by anterior and posterior approach. Although this technique is effective, it has a lot of disadvantages. So investigators introduce another surgical technique.

DETAILED DESCRIPTION:
Although hemivertebra resection technique can obtain satisfactory clinical outcome, it has its disadvantages. Because of the presence of vertebral arteries, the procedure of cervical hemivertebra resection is not only difficult and risky, but also time and labor consuming. The operation is a great challenge to the skill, physical strength and energy of the surgical team. Meanwhile, hemivertebra resection and compression on convex side may lead to iatrogenic foraminal stenosis and increase the incidence of nerve root palsy at the corresponding segment after surgery. The shortening of the convex side may further aggravate the patient's existing short neck deformity, which is not conducive to the recovery of patient's appearance. Therefore, our department pioneer a new surgical technique to avoid hemivertebra resection in 2015, which is distraction and lateral opening on concave side. This technique extends the concave side through intervertebral space where the concave apex locates or adjacent intervertebral space to achieve the purpose of scoliosis correction. The avoidance of hemivertebra resection significantly reduces the difficulty and risk of the surgery. This procedure tries to make up for the patient's congenital anatomical deficiency and lengthen the concave side. Although there is no need to expose vertebral artery, preoperative CTA(computed tomography angiography) should be performed routinely to determine whether there is abnormality in vertebral artery and whether it will interfere with the distraction on concave side and the placement of prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* the presence of torticollis caused by congenital cervical scoliosis (defined as a Cobb angle of >10°)
* operation and follow-up were performed in our hospital

Exclusion Criteria:

* Patients with other causes of torticollis appearance, such as muscular torticollis, ocular torticollis, neurogenic torticollis, etc.
* Patients with other spinal deformity or disease, such as cervical kyphosis or kyphoscoliosis, congenital deformity of middle and lower thoracic vertebra, lumbar vertebra, ankylosing spondylitis, severe ossification of cervical posterior longitudinal ligament, etc.
* Cervical infectious diseases, cervical primary or metastatic tumor
* Have a history of spinal trauma or surgery
* Imaging data are incomplete or of poor quality.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with congenital cervical scoliosis were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
the structural Cobb angle | one week pre operation
  the large curve in the segments with vertebral deformities causing clinical asymmetry or head deviation and needs to be surgically corrected
the structural Cobb angle | one week after surgery
  the large curve in the segments with vertebral deformities causing clinical asymmetry or head deviation and needs to be surgically corrected
the structural Cobb angle | through study completion, an average of 1 year
  the large curve in the segments with vertebral deformities causing clinical asymmetry or head deviation and needs to be surgically corrected
distal compensatory Cobb angle | one week pre operation
  the small curve without vertebral deformities
distal compensatory Cobb angle | one week after surgery
  the small curve without vertebral deformities
distal compensatory Cobb angle | through study completion, an average of 1 year
  the small curve without vertebral deformities
mandibular incline | one week pre operation
  the angle between the horizontal line and the line through the mandibular angles on both sides
mandibular incline | one week after surgery
  the angle between the horizontal line and the line through the mandibular angles on both sides
mandibular incline | through study completion, an average of 1 year
  the angle between the horizontal line and the line through the mandibular angles on both sides
clavicle angle | one week pre operation
  the angle between the horizontal line and the line through the clavicular distal end on both sides
clavicle angle | one week after surgery
  the angle between the horizontal line and the line through the clavicular distal end on both sides
clavicle angle | through study completion, an average of 1 year
  the angle between the horizontal line and the line through the clavicular distal end on both sides

SECONDARY OUTCOMES:
blood loss | during operation
  blood loss during operation
surgical time duration | during operation
  surgical time duration during operation
complications | peroperative period
  complications during and after operation

CONTACTS AND LOCATIONS:
Overall Officials: Yu Sun, MD, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No